CLINICAL TRIAL: NCT05535621
Title: 68Ga-HER2 Affibody PET/CT Imaging for HER2-Positive Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xiaohua Zhu, Professor, Tongji Hospital
Other Study IDs: TJ-IRB20211129
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: HER2-Positive Cancer
Keywords: HER2; PET

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of HER2 alterations in pan-cancer indicates a broader range of application of HER2-targeted therapies. immunohistochemistry (IHC) or amplification by fluorescence in situ hybridization (FISH) is currently the most commonly used method for evaluation of HER-2 status in cancer patients. However, biopsies are spatiotemporally limited because of the highly heterogeneous expression of HER2. Patients with false-negative HER2 results may miss the chance for targeted therapy. Additionally, the HER2 status can change during the disease process.

A investigational imaging tracer named 68Ga-HER2 Affibody binds to HER-2 receptors. Previous studies in human have shown the efficacy of 68Ga-HER2 Affibody in detecting HER2 positive breast cancer and gastric cancer without any observed toxicity. However, studies are still insufficient and limited to breast cancer and gastric cancer.

The investigators hypothesized that 68Ga-HER2 Affibody PET imaging can noninvasively assess HER2 status in metastatic or recurrent solid tumors including breast cancer, gastrointestinal tumors, head and neck squamous tumors, bladder cancer, lung cancer and uterine tumors lesion. In this study, efficacy of 68Ga-HER2 Affibody in detecting HER2 positive cancer lesions and change of patient management based on 68Ga-HER2 Affibody PET will be determined.

DETAILED DESCRIPTION:
The prevalence of HER2 alterations in pan-cancer indicates a broader range of application of HER2-targeted therapies. Tumors including breast cancer, gastrointestinal tumors, head and neck squamous tumors, bladder cancer, lung cancer and uterine tumors exhibited high HER2 indices together with HER2 amplification or overexpression, which may benefit from HER2-targeted therapies.

immunohistochemistry (IHC) or amplification by fluorescence in situ hybridization (FISH) is currently the most commonly used method for evaluation of HER-2 status in cancer patients. However, biopsies are spatiotemporally limited because of the highly heterogeneous expression of HER2. Patients with false-negative HER2 results may miss the chance for targeted therapy. Additionally, the HER2 status can change during the disease process.

A investigational imaging tracer named 68Ga-HER2 Affibody binds to HER-2 receptors. Previous studies in human have shown the efficacy of 68Ga-HER2 Affibody in detecting HER2 positive breast cancer and gastric cancer without any observed toxicity. However, studies are still insufficient and limited to breast cancer and gastric cancer.

The investigators hypothesized that 68Ga-HER2 Affibody PET imaging can noninvasively assess HER2 status in metastatic or recurrent solid tumors including breast cancer, gastrointestinal tumors, head and neck squamous tumors, bladder cancer, lung cancer and uterine tumors lesion. In this study, efficacy of 68Ga-HER2 Affibody in detecting HER2 positive cancer lesions and change of patient management based on 68Ga-HER2 Affibody PET will be determined.

ELIGIBILITY:
Inclusion Criteria:

patients with clinically diagnosed HER2-Positive tumor subjects need to sign the informed consent

Exclusion Criteria:

* Pregnant women; renal failure (serum Cr>3mg/dl); Patients with claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HER2-Positive tumor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 1 year
  SUVmax

CONTACTS AND LOCATIONS:
Overall Officials: ZHU XIAOHUA, DR, Principal Investigator — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zou S, Liu Z, Zhou J, Song S, Wang D, Zhu D, Cheng S, Cheng Z, Zhu Y, Yu T, Pan D, Yang M, Zhu X. Non-invasive assessment of HER2 expression in patients with urothelial carcinoma using [68Ga]Ga-HER2 affibody PET/CT imaging: preliminary clinical findings. Eur J Nucl Med Mol Imaging. 2025 Jul;52(8):2782-2791. doi: 10.1007/s00259-025-07142-0. Epub 2025 Feb 14. PMID 39951137